CLINICAL TRIAL: NCT06945354
Title: Intra Oral Scan and CBCT Aided Diagnosis of Dental Plaque and Caries
Status: Not yet recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0383
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries (Diagnosis); Dental Plaque (Diagnosis)
MeSH Terms: conditions — Dental Caries; Disease; Dental Plaque

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- caries diagnosis visual and bitewing: caries diagnosis intra oral scan and bitewing
- caries diagnosis CBCT: take a CBCT and registration caries
- Intra oral scan and bitewing: An intra-oral scan and bitewings are taken and 2 weeks later, caries is registered on the basis of this intra oral scan and bitewings
- plaque visual: registration plaque with visuals
- plaque color record visual: registration with plaque color record
- plaque Intra oral scan: registration plaque with intra-oral scan
- plaque color record with Intra-oral scan: registration plaque color record with intra-oral scan
- caries diagnosis fluorescence: registration caries with fluorescence of intra-oral scan

SUMMARY:
In this prospective controlled trial, patients will be enrolled at the University Hospital Ghent. Inclusion criteria are: age between 18 and 70 years old, presence of 20 or more teeth, and have a minimum one carious tooth surface. All participants have to sign an informed consent. Pregnant women will be excluded. First an intra-oral scan will be taken for visual plaque detection. Thereafter, plaque scores will be noted after visual inspection and with plaque staining. After supra-gingival calculus removal and oral hygiene instructions bite-wing radiographs will be taken and a visual caries inspection will be performed. Finally, a new intra-oral scan will be taken for visual caries detection, followed by a CBCT scan.

Minimally 2 weeks after this intervention, plaque-scores and caries-scores will be measured by an independent researcher and the same researcher on the intra-oral scans, CBCT and radiographs(Pictures taken with X-rays to view the inside of your teeth and jawbone)(for caries detection).

The following variables will be measured:

1. Plaque measurement: 1) Plaque detection using intra-oral scan images (white light (and fluorescence)) will be performed and compared with 2) the assessment of visual plaque detection and 3) using plaque staining (golden standard). The findings will be recorded in a plaque status through the website www.parodontalstatus. And exported to be attached to the anonymized patient file.
2. Caries: The results of caries detection by intra-oral scan and bite-wing radiographs will be compared with the results of clinical caries detection and bite-wing radiographs on one hand and the CBCT images on the other hand. ICDAS scores will be registered for the visual assessment, CBCT and bite-wing radiograph images assessment.

The following step-by-step protocol will be used:

The digital data, including images, that will be the subject of the research will be acquired using 3SHAPE's Trios 5 intra-oral scan. The CBCT image will be made with the ProMax 3D of Planmeca. These two imaging techniques will be the only study specific handeling during the study.

1. explanation to patients
2. take an intra-oral scan (STUDY SPECIFIC)
3. conventional visual inspection and palpation plaque scoring
4. plaque staining (record with parostatus.ch)
5. take an intra-oral scan with plaque staining in a situation that is viewed on site, in the mouth, without removing or moving anything.(STUDY SPECIFIC)
6. calculus removal and cleaning
7. take bite-wing radiographs
8. visual caries detection
9. take a thirth intra-oral scan (STUDY SPECIFIC)
10. CBCT scan (STUDY SPECIFIC)
11. plaque detection on IOS images and caries detection using IOS images and CBCT images

ELIGIBILITY:
Inclusion Criteria:age between 18 and 70 years old, presence of 20 or more teeth, and have a minimum one carious tooth surface -

Exclusion Criteria:Pregnant women will be excluded -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population is selected from Ghent university hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
caries diagnosis | one time measurement ( visual inspection ) 2weeks later, inspection of intra-oral scan and CBCT
  sensitivity specificity and area-under-curve values will be determined using receiver operating characteristic curve analysis
plaque diagnosis | one time measurement ( visual inspection) and 2 weeks later inspection of intra-oral scan and 2 weeks
  sensitivity specificity and area-under-curve values will be determined using receiver operating characteristic curve analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent university hospital, Ghent, Gent, Belgium

IPD SHARING:
Plan to Share IPD: No